CLINICAL TRIAL: NCT00275184
Title: A Randomised Study of the Optimal Bowel Preparation for Routine Capsule Endoscopy Using Citramag and Senna or Metoclopramide
Brief Title: Bowel Preparation and Prokinetics in Capsule Endoscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 05/CE/94; REC 05/Q0405/94; EudraCT No: 2005-004423-19
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Small Bowel Disease; Gastrointestinal Hemorrhage; Refractory Anemia
Keywords: Bowel preparation; capsule endoscopy; randomised; Citramag; Senna; Metoclopramide; Patients referred for Capsule endoscopy; occult/overt gastrointestinal bleeding; other suspected small bowel pathology
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Anemia, Refractory | interventions — Sennosides; Metoclopramide

INTERVENTIONS:
Drug: Senna
Drug: Citramag powder
Drug: Metoclopramide

SUMMARY:
The aim of this study is to determine whether taking bowel preparation (citramag and senna) or a medicine to speed up transit through the stomach (metoclopramide), will improve the quality of the images seen, increase the transit through the small bowel, and increase the rate of completion of capsule endoscopy.

The secondary objective is to determine whether patients could routinely tolerate this bowel preparation prior to capsule endoscopy and whether the diagnostic yield of capsule endoscopy is improved.

DETAILED DESCRIPTION:
Capsule endoscopy is a diagnostic tool for the detection of small bowel disease allowing noninvasive endoscopic examination of the entire small bowel without the need for sedation. Its limited battery life of 8+/-1 hours means it is paramount that the Capsule reaches the caecum, visualizing the whole of the small intestine, and also that the mucosal views obtained are clear, facilitating detection of pathologic lesions.

So far no optimal protocol for bowel preparation prior to Capsule endoscopy has been established. Recently, several studies have shown that bowel preparation with polyethylene glycol significantly reduces both gastric and small bowel transit times. Similarly, visualization of the small intestine and therefore 'diagnostic yield' have both been shown to be improved by both sodium phosphate and polyethylene glycol preparation. A more recent study by Selby et al also demonstrates that the prokinetic agent metoclopramide (which is known to promote emptying of the stomach) reduced both stomach and small bowel transit time, increasing completion rates from 76% to 97%).

The proposal is to perform a randomised, controlled study using Citramag and Senna bowel preparation or Metoclopramide to determine whether test completion rates are improved and whether the images of the bowel are of better quality.

The hypothesis is that the improved wall visibility and increased completion rates will improve the diagnostic yield of Capsule endoscopy and therefore improve patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 who have been referred for capsule endoscopy

Exclusion Criteria:

* Under 18
* Known or suspected gastrointestinal tract obstruction as this may impede passage of the capsule
* Known small bowel stricture or fistula as this may impede capsule passage
* Pregnancy, breast feeding or phaeochromocytoma as metoclopramide is contraindicated
* Recent gastrointestinal surgery in view of the risk of impeded capsule passage
* Permanent cardiac pacemaker or implantable defibrillator in-situ to avoid the risk of possible interference
* Congestive cardiac failure as citramag is contraindicated in such patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-01

PRIMARY OUTCOMES:
Quality of capsule endoscopic images, stomach and small bowel transit times and capsule completion rates to the end of the small bowel

SECONDARY OUTCOMES:
The tolerance of the bowel preparation to indicate future usage

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Fraser, MB BCH, MD, FRCP, Principal Investigator — St Mark's Hospital, North West London Hospitals NHS Trust
Locations (1):
- St Mark's Hospital, North West London Hospitals NHS Trust, London, United Kingdom